CLINICAL TRIAL: NCT02983240
Title: Electrical Inhibition (EI): A Preliminary Study to Prevent the Uterine Contractions of Human Preterm Labor and Preterm Birth
Brief Title: Electrical Inhibition of Human Preterm Contractions
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: PI change
Sponsor: e-Bio Corp (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB201601699 - A; OCR26522 (Other: UF OnCore); E-BIO CORP (Other: PRO00038898)
Record Dates: First submitted 2016-12-02; First posted 2016-12-06 (Estimated); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Preterm Labor; PreTerm Birth; Preterm Labor With Delivery Nos
MeSH Terms: conditions — Obstetric Labor, Premature; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- 60 Minute Study (Experimental): After a 20-minute pre-intervention control period the electrical inhibition will be used intermittently, only when there is monitored contraction, during the 20-minute intervention study period. At the end of the intervention period there will be a 20-minute post-intervention control period. The FHR patterns, tocogram, EMG and EHG, and fECG recordings will be compared to before and after the use of the electrical uterine pacemaker device.
  Interventions: Device: Electrical Uterine Pacemaker
- 80 Minute Study (Experimental): After a 20-minute pre-intervention control period the electrical inhibition will be used intermittently, only when there is monitored contraction, during the 40-minute intervention study period. At the end of the intervention period there will be a 20-minute post-intervention control period. The FHR patterns, tocogram, EMG and EHG, and fECG recordings will be compared to before and after the use of the electrical uterine pacemaker device.
  Interventions: Device: Electrical Uterine Pacemaker
- 120 Minute Study (Experimental): After a 20-minute pre-intervention control period the electrical inhibition will be used intermittently, only when there is monitored contraction, during the 80-minute intervention study period. At the end of the intervention period there will be a 20-minute post-intervention control period. The FHR patterns, tocogram, EMG and EHG, and fECG recordings will be compared to before and after the use of the electrical uterine pacemaker device.
  Interventions: Device: Electrical Uterine Pacemaker

INTERVENTIONS:
Device: Electrical Uterine Pacemaker — The catheter is placed under ultrasound guidance into the posterior vaginal fornix next to the external cervical os. The electrode connectors are attached to the EI device. Activating the EI device involves: 1) turning the current pulse duration rotary dial clockwise to the desired setting; this is an important setting and should be set at 20ms; 2) turning the current frequency rotary dial clockwise to the desired setting; 3) turn on the EI device on with the on/off toggle switch; 4) SLOWLY turning the current strength rotary dial clockwise to the desired setting, at this time the red light should be flashing. Usually 5-10mA of current is sufficient, but 20 mA is a maximum. Based on the tocometer recordings the least amount of EI current is given to inhibit the uterine contractions.

SUMMARY:
The purpose of this study is to explore a new method to stop preterm uterine contractions using an electrical device. The device, an "electrical pacemaker for the uterus," has been approved by the Food and Drug Administration (FDA) for clinical research in pregnant women. The purpose of this study is to evaluate the feasibility and safety of the device. The investigators hypothesize that human preterm uterine contractions can be safely and objectively inhibited with a weak electrical current provided by an electrical inhibition (EI)/uterine pacemaker device, and that this effect relates to the timing and length of EI exposure.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effectiveness of a new method of preventing the human preterm uterine contractions of labor during electrical monitoring. The objective is to test a method for the inhibition of human preterm uterine contractions with an electrical pacemaker, electrical inhibition (EI). The study will investigate EI associated changes in preterm uterine contraction frequency as monitored by objective uterine tocodynamometry and adjunct electromyography (EMG) and electrohysterogram (EHG). The endpoint is the statistically significant EI induced decrease in the gold standard tocodynamometric monitored preterm uterine contraction frequency. The adjunct EMG and EHG monitoring provides valuable adjunct data about the electrical activity of the preterm uterine contractions and the effect of EI on this activity.

The investigators hypothesize that human preterm uterine contractions can be safely and objectively inhibited with a weak electrical current provided by an electrical inhibition (EI)/uterine pacemaker device. This effect can be assessed by the use of a non-invasive tocodynamometer. It has been previously been shown that the frequency of contractions during preterm labor can be lowered by EI applied by the use of an intravaginal catheter carrying electrodes similar to a cardiac pacemaker (Karsdon et al). The investigators hypothesize that this effect relates to the timing and length of EI exposure.

ELIGIBILITY:
Inclusion Criteria:

* Wong-Baker pain score ≤ 6
* Pregnancy Depression Scale score < 16
* Informed consent form signed and dated by patient
* Be willing and able to comply with study requirements
* Be between 18-50 years of age
* Be between 23 to 36 5/7 weeks pregnant with a singleton gestation
* Cervical dilation of ≤ 6 cm
* A normal spontaneous vaginal delivery (NSVD) expected
* Suspected to have preterm labor, as defined by the American College of Obstetricians and Gynecologists and the American Academy of Pediatrics, as follows.78

  * Persistent uterine contractions (4 every 20 minutes, or 8 every 60 minutes)
  * And any one or more of the following:
  * Documented cervical change
  * 1 cm cervical dilatation and progressing

    -> 80% cervical effacement
  * Be admitted to the maternity unit with the diagnosis of preterm labor or preterm contractions

Exclusion Criteria:

* Severe preeclampsia
* Severe abruption placenta
* Abnormal placentation (i.e. placenta previa)
* Rupture of amniotic membranes
* Active preterm labor with cervical dilation > 6 cm
* Exposed amniotic membranes
* Vaginal bleeding > 10 cc
* Frank chorioamnionitis
* Fetal death
* Fetal anomaly incompatible with life
* Severe fetal growth restriction (EFW < 5%)
* Uterine anomalies (i.e. bicornuate uterus, uterine didelphys)
* Mature fetal lung studies
* Maternal cardiac arrhythmias
* HIV, Hepatitis C, Hepatitis B
* History of herpes simplex virus (HSV)
* A permanent cardiac pacemaker
* A fetal cardiac arrhythmia
* Contraindication for tocolysis e.g. premature rupture of the amniotic membranes allowing for ascending intrauterine infection with group B streptococcus or GBS (beta hemolytic streptococcus, S. agalactiae) or other micro-organisms.
* IV or po narcotic pain medication < 12 hours prior to admission (regional anesthesia, long acting oral maintenance opiates i.e. methadone, Suboxone, Subutex not included in exclusion criteria)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2026-01-21 (Estimated); Study Completion 2026-01-21 (Estimated)

PRIMARY OUTCOMES:
Uterine contraction frequency during labor as measured by external uterine tocodynamometric monitoring | Change from 20, 40, and 80 minutes

SECONDARY OUTCOMES:
FHR pattern as measured by the maternal-fetal monitor | Change from 60 and 120 minutes
EMG monitoring as measured by LaborView Device | Change from 60 and 120 minutes
EHG monitoring as measured by LaborView Device | Change from 60 and 120 minutes
fECG monitoring as measured by LaborView Device | Change from 60 and 120 minutes
Maternal pain medication administration | Before and after use of electrical uterine pacemaker, assessed up to 120 minutes
Maternal heart rate | Change from 60 and 120 minutes

OTHER OUTCOMES:
Adverse events | Before and after use of electrical uterine pacemaker, assessed up to 120 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Karsdon, MD, Study Chair — New York University Lagone Medical Center; John Smulian, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karsdon J, El Daouk M, Huang WM, Ashmead GG. Electrical pacemaker as a safe and feasible method for decreasing the uterine contractions of human preterm labor. J Perinat Med. 2012 Nov;40(6):697-700. doi: 10.1515/jpm-2012-0136. PMID 23089601